CLINICAL TRIAL: NCT03001271
Title: Acute Effect of Agiotensin-(1-7) on Bood Pressure and Heart Rate in Healthy and Hypertensive Subjects
Brief Title: Acute Effect of Agiotensin-(1-7) in Healthy and Hypertensive Subjects
Acronym: Ang-(1-7)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 4576/10
Record Dates: First submitted 2016-12-02; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Hypertension
Keywords: Angiotensin-(1-7); Renin-angiotensin System; Autonomic Nervous System
MeSH Terms: conditions — Hypertension | interventions — angiotensin I (1-7)

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Healthy Subjects (Experimental): Placebo and Angiotensin-(1-7) acute infusion
  Interventions: Drug: Angiotensin 1-7; Other: Placebo
- Hypertensive Subjects (Experimental): Placebo and Angiotensin-(1-7) acute infusion
  Interventions: Drug: Angiotensin 1-7; Other: Placebo

INTERVENTIONS:
Drug: Angiotensin 1-7
  Other Names: Angio-1-7
Other: Placebo

SUMMARY:
In the modern concept of Renin-angiotensin System, Angiotensin-(1-7) plays a key role and demonstrates promising therapeutic potential due to it is generally opposite effects to Angiotensin II. The aim is to evaluate the effect of Ang-(1-7) acute administration on systolic and diastolic blood pressure (SBP and DBP) and heart rate (HR) in healthy and hypertensive subjects.

ELIGIBILITY:
Healthy Group Inclusion Criteria:

* arterial pressure <140/90 mmHg
* body mass index (BMI) between 18,5 and 29 Kg/m2

Hypertensive Group Inclusion Criteria:

* anti-hypertensive drug treatment
* ambulatory blood pressure monitoring (ABMP) >130/85 mmHg
* body mass index between 18,5 and 29 Kg/m2

Healthy Group Exclusion Criteria:

* drug treatment
* recent surgeries
* pregnancy
* previous cardiovascular events
* high performance athletes
* dislipidemia
* diabetes
* renal injury
* obesity (BMI above 30 kg/m2)
* alcoholism
* smoking.

Hypertensive Group Exclusion Criteria:

* recent surgeries
* pregnancy
* beta-blockers drug treatment
* previous cardiovascular events
* high performance athletes
* dislipidemia
* diabetes
* renal injury
* obesity (BMI above 30 kg/m2)
* alcoholism
* smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Absence of adverse effects after Ang-(1-7) acute administration | Along 25 hours

SECONDARY OUTCOMES:
Blood Pressure Changes after Ang-(1-7) administration | Recording along 24 hours
  absence of measure changes in blood pressure or heart rate (increase or decrease)
Ang-(1-7) effects on Blood Pressure Variability | Along 1 hours after Ang-(1-7) acute administration
  Response of autonomic nervous system, registered for 1 hours, after Ang-(1-7) acute administration
Heart Rate Changes after Ang-(1-7) administration | Recording along 24 hours
Ang-(1-7) effects on Heart Rate Variability | Along 1 hours after Ang-(1-7) acute administration
  Response of autonomic nervous system, registered for 1 hours, after Ang-(1-7) acute administration